CLINICAL TRIAL: NCT06778317
Title: Evaluation of the Circulating Epigenetic Biomarker MSEPT9 for Predicting the Occurrence of Hepatocellular Carcinoma in Patients with Cirrhosis: a Prospective Multicenter Trial (SEPT9_SuRV)
Brief Title: MSEPT9 Biomarker for Predicting Hepatocellular Carcinoma Occurrence in Patients with Cirrhosis
Acronym: SEPT9_SuRV
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: New Day Diagnostics (Network)
Responsible Party: Sponsor
Other Study IDs: 2022-A01664-39
Record Dates: First submitted 2024-12-27; First posted 2025-01-16 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-12

CONDITIONS: Hepatocellular Carcinoma (HCC); Cirrhosis; Risk Prediction for Liver Cancer; Epigenomics
Keywords: Hepatocellular Carcinoma; Cirrhosis; mSEPT9 Biomarker; Epigenetics; Risk Prediction; Liver Cancer Surveillance; Prospective Cohort Study; Non-Invasive Biomarkers; Personalized Medicine; Epigenomics; Risk Stratification
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The biospecimens retained in this study include plasma samples and genetic material (DNA) collected from patients with cirrhosis during routine blood draws at each of the 11 scheduled visits (baseline and every 6 months for 60 months). For each visit, two 10 mL blood samples will be collected in EDTA tubes. Plasma will be extracted, aliquoted, and stored at -80°C for subsequent analysis of the mSEPT9 epigenetic biomarker.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients With Cirrhosis Without Hepatocellular Carcinoma at Baseline: This cohort includes 400 patients with cirrhosis who do not have hepatocellular carcinoma (HCC) at the time of inclusion. Participants will undergo standard clinical, biological, and radiological evaluations every six months for a total follow-up duration of 60 months, in accordance with international guidelines for cirrhosis management. In addition to routine assessments, blood samples will be collected at each visit for the analysis of the circulating epigenetic biomarker mSEPT9. This biomarker will be tested to evaluate its utility in predicting the occurrence of HCC during the follow-up period. The results of the mSEPT9 test will not influence clinical management during the study.
  Interventions: Diagnostic Test: Circulating mSEPT9 Biomarker Testing

INTERVENTIONS:
Diagnostic Test: Circulating mSEPT9 Biomarker Testing — This intervention involves the analysis of the circulating epigenetic biomarker mSEPT9 through plasma samples collected from patients with cirrhosis. The mSEPT9 test evaluates the methylation status of the SEPT9 gene promoter using a triplicate assay. A "switch" in the test status, defined as a transition from triple-negative (no methylation detected in any triplicate) to at least one positive triplicate, is being investigated as a prognostic marker for the development of hepatocellular carcinoma (HCC).
  The mSEPT9 test is conducted on plasma samples collected during routine blood draws at each of the 11 scheduled study visits. Samples are processed and analyzed in batches using specialized high-throughput equipment provided by Epigenomics/New Day Diagnostics. Results of the mSEPT9 test are not shared with clinicians during the study period to avoid influencing patient management, ensuring the test is purely investigational in this context.
  Other Names: Plasma mSEPT9 Testing; Epigenetic Biomarker Analysis; mSEPT9 Methylation Test

SUMMARY:
This study aims to evaluate the role of the circulating epigenetic biomarker mSEPT9 in predicting the risk of hepatocellular carcinoma (HCC) in patients with cirrhosis. HCC is a primary liver cancer that frequently develops in individuals with cirrhosis, and early detection is critical for improving outcomes. This research involves 400 patients with cirrhosis who will be followed every six months for up to 60 months. During these visits, blood samples will be collected to analyze mSEPT9 levels. By identifying changes in this biomarker, the study seeks to improve early diagnosis and personalize surveillance strategies, potentially enhancing patient survival and quality of life.

DETAILED DESCRIPTION:
This study is a prospective, multicenter cohort trial designed to assess the prognostic utility of the circulating epigenetic biomarker mSEPT9 in predicting the development of hepatocellular carcinoma (HCC) among patients with cirrhosis. The trial involves 400 participants who are confirmed to have cirrhosis and no evidence of HCC at baseline.

The study's primary focus is to evaluate the association between a "switch" in the mSEPT9 test-from a triple-negative status (no methylation detected across triplicate assays) to at least one positive triplicate-and the subsequent occurrence of HCC. Secondary objectives include assessing this association across different etiologies of cirrhosis (e.g., viral hepatitis, alcohol-related liver disease, nonalcoholic steatohepatitis) and its correlation with HCC-related mortality.

Participants will undergo standardized clinical, biological, and imaging assessments every six months over a follow-up period of 60 months, as per international guidelines for cirrhosis management. In addition to routine care, blood samples will be collected at each visit for mSEPT9 testing. These samples will be processed, stored at -80°C, and analyzed in batches to assess mSEPT9 levels.

The findings from this study are expected to address the unmet need for reliable, non-invasive biomarkers for HCC risk prediction, potentially leading to personalized surveillance strategies and earlier intervention for patients with cirrhosis. Data will be managed using an electronic case report form (eCRF) to ensure secure, standardized documentation across all participating centers. Results from mSEPT9 testing will not influence clinical management during the study period but will be analyzed to determine their predictive value for HCC development and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Patients diagnosed with cirrhosis confirmed by clinical, biochemical, radiological, or histological criteria.
* Cirrhosis attributable to one or more of the following etiologies: alcohol, hepatitis C (HCV), hepatitis B (HBV), nonalcoholic steatohepatitis (NASH), hemochromatosis, autoimmune hepatitis, primary biliary cholangitis, primary sclerosing cholangitis, or cryptogenic causes.
* Patients actively followed in one of the participating study centers.
* Patients affiliated with a social security program or equivalent.
* Patients with a body weight greater than 45 kg.
* Patients who have been fully informed about the study procedures and have provided oral informed consent.

Exclusion Criteria:

* History of hepatocellular carcinoma (HCC).
* History of any other primary or secondary malignant liver tumor.
* Diagnosis of malignancy or hematologic disorders within the past 5 years (without time limitation for hematologic malignancies).
* Patients currently undergoing hemodialysis.
* Pregnant or breastfeeding women.
* Individuals under legal protection (e.g., guardianship, curatorship) or unable to provide consent.
* Minors or individuals younger than 18 years.
* Individuals deprived of liberty by judicial or administrative order.
* Patients with psychiatric conditions receiving care under legal constraints (e.g., articles L.3212-1 and L.3213-1).
* Patients unable to comply with the study protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of 400 adult patients with confirmed cirrhosis who are actively followed in specialized hepatology centers across multiple institutions. Participants must not have hepatocellular carcinoma (HCC) at the time of enrollment and must meet specific inclusion criteria, including established cirrhosis etiology and eligibility for routine clinical follow-up. Patients with conditions that may interfere with the study objectives, such as a history of malignancy or ongoing hemodialysis, are excluded. This cohort represents a diverse range of cirrhosis etiologies, including viral hepatitis, alcohol-related liver disease, and nonalcoholic steatohepatitis (NASH), to ensure the generalizability of findings.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-03-03 (Estimated); Primary Completion 2030-03-04 (Estimated); Study Completion 2031-03-03 (Estimated)

PRIMARY OUTCOMES:
Association Between mSEPT9 Test Switch and Hepatocellular Carcinoma (HCC) Development | Annually for up to 60 months or until the occurrence of HCC, whichever occurs first.
  Evaluate the relationship between a 'switch' in the mSEPT9 test result-defined as a transition from triple-negative (no methylation detected across all triplicates) to at least one positive triplicate-and the occurrence of hepatocellular carcinoma (HCC), as diagnosed using international criteria established by the AASLD.

SECONDARY OUTCOMES:
Association Between mSEPT9 Test Switch and HCC Development by Cirrhosis Etiology | Annually for up to 60 months or until the occurrence of HCC, whichever occurs first.
  Assess the association between a 'switch' in mSEPT9 test results and the development of hepatocellular carcinoma (HCC), as diagnosed using international criteria (AASLD), across subgroups categorized by cirrhosis etiology, including alcohol use, hepatitis B (HBV), hepatitis C (HCV), and nonalcoholic steatohepatitis (NASH). A 'switch' in the mSEPT9 test result is defined as a transition from triple-negative (no methylation detected across all triplicates) to at least one positive triplicate.
Association Between mSEPT9 Test Results and HCC-Related Mortality | Annually for up to 60 months or until HCC-specific death occurs.
  HCC-specific mortality, defined as death attributable to hepatocellular carcinoma based on international classification of diseases (ICD) coding and/or clinical determination, stratified by positive or negative mSEPT9 test results (performed in triplicate).
Establishment of a Biobank for Genomic and Epigenomic Analysis | For each participant, samples will be collected at enrollment (baseline) and during follow-up visits every 6 months for up to 60 months.
  Number of Plasma and DNA Samples Collected and Stored for Genomic and Epigenomic Analysis, Including Data on Sample Quality, Quantity.

CONTACTS AND LOCATIONS:
Overall Officials: Mr. Franck Schreiner, Study Director — Regional and University Hospital Center of Nancy
Locations (1):
- Regional and University Hospital Center of Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Yes
The study will share individual participant data (IPD) related to anonymized clinical, biological, and imaging results, as well as the results of mSEPT9 biomarker analyses.
  This includes:
  * Demographic data
  * Clinical characteristics, including cirrhosis etiology and disease severity (e.g., Child-Pugh score)
  * Results from routine imaging and biological assessments
  * mSEPT9 test results (e.g., triple-negative, positive status)
  * Outcome measures, such as the occurrence of hepatocellular carcinoma (HCC) and mortality
  All shared data will be pseudo-anonymized to ensure participant confidentiality and will be accessible to researchers upon reasonable request, in accordance with regulatory and ethical guidelines.
Supporting Information: Study Protocol, SAP, Analytic Code
Access Criteria: The individual participant data (IPD) and supporting information will be available starting 12 months after the publication of the study results. IPD related to outcomes outside the primary and secondary objectives of the study may be discussed and shared on a case-by-case basis, contingent on appropriate approvals and compliance with applicable regulations.

REFERENCES:
- [Background] Oussalah A, Rischer S, Bensenane M, Conroy G, Filhine-Tresarrieu P, Debard R, Forest-Tramoy D, Josse T, Reinicke D, Garcia M, Luc A, Baumann C, Ayav A, Laurent V, Hollenbach M, Ripoll C, Gueant-Rodriguez RM, Namour F, Zipprich A, Fleischhacker M, Bronowicki JP, Gueant JL. Plasma mSEPT9: A Novel Circulating Cell-free DNA-Based Epigenetic Biomarker to Diagnose Hepatocellular Carcinoma. EBioMedicine. 2018 Apr;30:138-147. doi: 10.1016/j.ebiom.2018.03.029. Epub 2018 Mar 28. PMID 29627389
- [Background] Nahon P, Layese R, Bourcier V, Cagnot C, Marcellin P, Guyader D, Pol S, Larrey D, De Ledinghen V, Ouzan D, Zoulim F, Roulot D, Tran A, Bronowicki JP, Zarski JP, Riachi G, Cales P, Peron JM, Alric L, Bourliere M, Mathurin P, Blanc JF, Abergel A, Serfaty L, Mallat A, Grange JD, Attali P, Bacq Y, Wartelle C, Dao T, Thabut D, Pilette C, Silvain C, Christidis C, Nguyen-Khac E, Bernard-Chabert B, Zucman D, Di Martino V, Sutton A, Roudot-Thoraval F, Audureau E; ANRS CO12 CirVir Group. Incidence of Hepatocellular Carcinoma After Direct Antiviral Therapy for HCV in Patients With Cirrhosis Included in Surveillance Programs. Gastroenterology. 2018 Nov;155(5):1436-1450.e6. doi: 10.1053/j.gastro.2018.07.015. Epub 2018 Jul 19. PMID 30031138
- [Background] Moon AM, Weiss NS, Beste LA, Su F, Ho SB, Jin GY, Lowy E, Berry K, Ioannou GN. No Association Between Screening for Hepatocellular Carcinoma and Reduced Cancer-Related Mortality in Patients With Cirrhosis. Gastroenterology. 2018 Oct;155(4):1128-1139.e6. doi: 10.1053/j.gastro.2018.06.079. Epub 2018 Jul 5. PMID 29981779
- [Background] Heimbach JK, Kulik LM, Finn RS, Sirlin CB, Abecassis MM, Roberts LR, Zhu AX, Murad MH, Marrero JA. AASLD guidelines for the treatment of hepatocellular carcinoma. Hepatology. 2018 Jan;67(1):358-380. doi: 10.1002/hep.29086. No abstract available. PMID 28130846
- [Background] Forner A, Reig M, Bruix J. Hepatocellular carcinoma. Lancet. 2018 Mar 31;391(10127):1301-1314. doi: 10.1016/S0140-6736(18)30010-2. Epub 2018 Jan 5. PMID 29307467
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: Management of hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):182-236. doi: 10.1016/j.jhep.2018.03.019. Epub 2018 Apr 5. No abstract available. Erratum In: J Hepatol. 2019 Apr;70(4):817. doi: 10.1016/j.jhep.2019.01.020. PMID 29628281
- [Background] Sharma SA, Kowgier M, Hansen BE, Brouwer WP, Maan R, Wong D, Shah H, Khalili K, Yim C, Heathcote EJ, Janssen HLA, Sherman M, Hirschfield GM, Feld JJ. Toronto HCC risk index: A validated scoring system to predict 10-year risk of HCC in patients with cirrhosis. J Hepatol. 2017 Aug 24:S0168-8278(17)32248-1. doi: 10.1016/j.jhep.2017.07.033. Online ahead of print. PMID 28844936
- [Background] Moran S, Martinez-Cardus A, Boussios S, Esteller M. Precision medicine based on epigenomics: the paradigm of carcinoma of unknown primary. Nat Rev Clin Oncol. 2017 Nov;14(11):682-694. doi: 10.1038/nrclinonc.2017.97. Epub 2017 Jul 4. PMID 28675165
- [Background] Hao X, Luo H, Krawczyk M, Wei W, Wang W, Wang J, Flagg K, Hou J, Zhang H, Yi S, Jafari M, Lin D, Chung C, Caughey BA, Li G, Dhar D, Shi W, Zheng L, Hou R, Zhu J, Zhao L, Fu X, Zhang E, Zhang C, Zhu JK, Karin M, Xu RH, Zhang K. DNA methylation markers for diagnosis and prognosis of common cancers. Proc Natl Acad Sci U S A. 2017 Jul 11;114(28):7414-7419. doi: 10.1073/pnas.1703577114. Epub 2017 Jun 26. PMID 28652331
- [Background] Ngwa JS, Cabral HJ, Cheng DM, Pencina MJ, Gagnon DR, LaValley MP, Cupples LA. A comparison of time dependent Cox regression, pooled logistic regression and cross sectional pooling with simulations and an application to the Framingham Heart Study. BMC Med Res Methodol. 2016 Nov 3;16(1):148. doi: 10.1186/s12874-016-0248-6. PMID 27809784
- [Background] Bruix J, Reig M, Sherman M. Evidence-Based Diagnosis, Staging, and Treatment of Patients With Hepatocellular Carcinoma. Gastroenterology. 2016 Apr;150(4):835-53. doi: 10.1053/j.gastro.2015.12.041. Epub 2016 Jan 12. PMID 26795574
- [Background] Villanueva A, Portela A, Sayols S, Battiston C, Hoshida Y, Mendez-Gonzalez J, Imbeaud S, Letouze E, Hernandez-Gea V, Cornella H, Pinyol R, Sole M, Fuster J, Zucman-Rossi J, Mazzaferro V, Esteller M, Llovet JM; HEPTROMIC Consortium. DNA methylation-based prognosis and epidrivers in hepatocellular carcinoma. Hepatology. 2015 Jun;61(6):1945-56. doi: 10.1002/hep.27732. Epub 2015 Mar 18. PMID 25645722
- [Background] Chaiteerakij R, Addissie BD, Roberts LR. Update on biomarkers of hepatocellular carcinoma. Clin Gastroenterol Hepatol. 2015 Feb;13(2):237-45. doi: 10.1016/j.cgh.2013.10.038. Epub 2013 Nov 23. PMID 24275343
- [Background] Mair RD, Valenzuela A, Ha NB, Ayoub WS, Daugherty T, Lutchman GA, Garcia G, Ahmed A, Nguyen MH. Incidence of hepatocellular carcinoma among US patients with cirrhosis of viral or nonviral etiologies. Clin Gastroenterol Hepatol. 2012 Dec;10(12):1412-7. doi: 10.1016/j.cgh.2012.08.011. Epub 2012 Aug 16. PMID 22902757
- [Background] Kakehashi A, Ishii N, Shibata T, Wei M, Okazaki E, Tachibana T, Fukushima S, Wanibuchi H. Mitochondrial prohibitins and septin 9 are implicated in the onset of rat hepatocarcinogenesis. Toxicol Sci. 2011 Jan;119(1):61-72. doi: 10.1093/toxsci/kfq307. Epub 2010 Oct 8. PMID 20935162
- [Background] El-Serag HB. Hepatocellular carcinoma. N Engl J Med. 2011 Sep 22;365(12):1118-27. doi: 10.1056/NEJMra1001683. No abstract available. PMID 21992124
- [Background] Bruix J, Sherman M; American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma: an update. Hepatology. 2011 Mar;53(3):1020-2. doi: 10.1002/hep.24199. No abstract available. PMID 21374666
- [Background] Berman K, Tandra S, Vuppalanchi R, Ghabril M, Sandrasegaran K, Nguyen J, Caffrey H, Liangpunsakul S, Lumeng L, Kwo P, Chalasani N. Hepatic and extrahepatic cancer in cirrhosis: a longitudinal cohort study. Am J Gastroenterol. 2011 May;106(5):899-906. doi: 10.1038/ajg.2010.477. Epub 2010 Dec 21. PMID 21179013
- [Background] deVos T, Tetzner R, Model F, Weiss G, Schuster M, Distler J, Steiger KV, Grutzmann R, Pilarsky C, Habermann JK, Fleshner PR, Oubre BM, Day R, Sledziewski AZ, Lofton-Day C. Circulating methylated SEPT9 DNA in plasma is a biomarker for colorectal cancer. Clin Chem. 2009 Jul;55(7):1337-46. doi: 10.1373/clinchem.2008.115808. Epub 2009 Apr 30. PMID 19406918
- [Background] Scott M, Hyland PL, McGregor G, Hillan KJ, Russell SE, Hall PA. Multimodality expression profiling shows SEPT9 to be overexpressed in a wide range of human tumours. Oncogene. 2005 Jul 7;24(29):4688-700. doi: 10.1038/sj.onc.1208574. PMID 15782116
- [Background] Boberg KM, Rocca G, Egeland T, Bergquist A, Broome U, Caballeria L, Chapman R, Hultcrantz R, Mitchell S, Pares A, Rosina F, Schrumpf E. Time-dependent Cox regression model is superior in prediction of prognosis in primary sclerosing cholangitis. Hepatology. 2002 Mar;35(3):652-7. doi: 10.1053/jhep.2002.31872. PMID 11870380